CLINICAL TRIAL: NCT05499156
Title: Safety of Injection of Placental Mesenchymal Stem Cell Derived Exosomes for Treatment of Resistant Perianal Fistula in Crohn's Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRCT20200413047063N3
Record Dates: First submitted 2022-05-30; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2021-09

CONDITIONS: Perianal Fistula in Patients With Crohn's Disease

STUDY DESIGN:
Intervention Model Description: This study includes two arms. The first one is the cases that are treated with MSC-derived exosomes and the controls do not receive exosomes and are treated with placebo
Who Masked: Participant, Outcomes Assessor
Masking Description: both the patient and the assessor are blind to the contents of injectibles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exosome therapy (Experimental): placenta-MSCs derived exosomes Exosomes are extracellular vesicles that are 30 to 150 nm in diameter. These vesicles are secreted from various cells. Mesenchymal stem cells exhibit immunomodulatory and anti-inflammatory properties by using paracrine effects. Exosomes, as a vehicle for signaling, are responsible for a significant part of cell-to-cell signaling. The preclinical animal studies manifested high safety and efficacy for MSC-derived exosome treatment on various fistulas and inflammatory bowel disease. In this study, we aimed to evaluate the safety and effectiveness of PlacentaMSCs derived exosomes in the treatment of patients with complex preanal fistula (Crohn's) in phases I and II of the clinical trial
  Interventions: Other: placenal MSC derived exosomes
- placebo (Experimental): placebo
  Interventions: Other: placenal MSC derived exosomes

INTERVENTIONS:
Other: placenal MSC derived exosomes — placenta-MSCs derived exosomes Exosomes are extracellular vesicles that are 30 to 150 nm in diameter. these vesicles are secreted from various cells. Mesenchymal stem cells exhibit immunomodulatory and anti- inflammatory properties by the use of paracrine effects. Exosomes as a vehicle for signaling, are responsible for a major part of cell to cell signaling. The preclinical animal studies manifested high safety and efficacy for MSC derived exosome treatment on various fistulas and inflammatory bowel disease. In this study we aimed to evaluate the safety and efficacy of PlacentaMSCs derived exosomes in treatment of patients with complex preanal fistula (non-crohn's) in phase I and II of clinical trial

SUMMARY:
Study aim:

Safety of Human Placenta Mesenchymal Stem Cells Derived Exosomes for treatment of perianal fistula in patients with Crohn's disease 2. Efficacy of Human Placenta Mesenchymal Stem Cells Derived Exosomes for treatment of refractory Anal Fistula in patients with Crohn's disease 3. Fistula changes in MRI studies, 12 weeks after treatment 4. Evaluation of quality of life in perianal fistula patient's questionnaire score before and 12 weeks after treatment

Participants/Inclusion and exclusion criteria:

inclusion criteria: 1. Age between 18-70 years old 2.Occurrence in patients with Crohn's disease 3. Informed consent Exclusion Criteria: 1. Active inflammatory bowel disease 2. Synchronous perianal abscess 3. Alcohol, narcotics and stimulant consumption 4. Having active Hepatitis B, C, HIV, or TB 5. Pregnancy and lactation 6.Uncontrolled diabetes mellitus 7. Evidence of surgical contraindication 8.Psychological disorders and noncooperative patient

Intervention groups:

Human Placenta Mesenchymal Stem Cells Derived Exosomes injected in fistula tract of patients with complex perianal Fistula in 3 weekly episodes, and it's safety and efficacy were evaluated.

Design:

this study includes two separate groups of cases and controls, each consisting of 40 participants randomly allocated for phase 2 of a clinical trial.

Settings and conduct:

Patients with complex perianal fistula referred to Imam Khomeini hospital will be included in the study if they contain inclusion criteria. The fistula was evaluated by clinical examination, and MRI and patients fill the quality of life questionnaire. Exosome injections are performed weekly for three consecutive weeks. Patients will be reexamined and fill out the questionnaire, and MRI will be done 12 weeks later. Recent findings will compare with the initial data. During this period, patients are examined for complications.

Main outcome variables:

Discharge amount; External orifice re-epithelialization; Inflammation, discharge and abscess larger than 2 cm in MR imaging; Quality of life questionnaire score, Inflammatory markers such as CRP, IL-6, TNF-a, calprotectin

DETAILED DESCRIPTION:
All patients who were enrolled in our study had refractory disease. These patients were previously treated and had unhealed cryptoglandular fistulas. The patients who were enrolled in this study were those who did not make any improvement after administration of 10 mg/kg of intravenous infliximab and seton placement. Patients were excluded if they had anti-TNF α treatment for less than six months, had no prior surgical interventions, or had a history of malignancies or immunodeficiency diseases. Pregnant patients were also excluded.

MSCs in third passage 3 were cultured in T175 flasks with D-MEM F12 culture medium (Gibco) supplemented with Pen/Strep, Strep, and 10 % exosome depleted FBS(Gibco) for 48 hours at 37 °C with a CO2 concentration of 5% at and humidity of 90 % humidity. Under 5% CO2. The conditioned media of MSCs (CM) were collected and centrifuged for 10 min at 400×g to eliminate suspended cells, 30 min at 2500×g to remove debris and apoptotic bodies, and then ultracentrifuged for 120 min at 100000×g (Beckman, USA). The supernatants were collected and further ultracentrifuged for 120 min at 100000×g. Then the pellets containing exosomes were dissolved in PBS.

To verify The production of MSC- derived exosomes, vesicle protein content was measured by Bradford colorimetric assay (BCA) from 100 ml of CM. The size distribution of MSC- derived exosomes were determined by dynamic light scattering (DLS). Moreover, to assess the expression of CD9, CD63 and CD81 were confirmed with flow cytometry and western blot., FITC mouse anti-CD63 (BD Pharmingen) and PE mouse anti-CD81 (BD Pharmingen) were used as reagents. Furthermore, the morphology and size of isolated exosomes were assessed using TEM by the previously set protocol in the previous study.

The procedure was undertaken in the operation room, and the patients were NPO 6 hours before the operation with intravenous sedation and oxygen supplementation with a mask. The patients, placed were placed in a lithotomy position. The external fistula opening was inspected, the tract was palpated, and using an Eisenhammer Retractor, the internal orifice was exposed seen. The lot was irrigated with saline several times using a small catheter to clear the pus and fecal material. After irrigation, a flexible fistula probe was inserted into the tract. Using the probe as a guide, we injected 5 mL of exosome solution into the tissue surrounding the lot. The injection depth was about 2about 2-3 mm of the soft tissue and sphincters of the anus. After the injection, the tract probe was extracted, the patients were under observation in the operation recovery rooming room recovery for 3 hours, and vital signs were monitored. The patients were then transferred to the surgery ward and were observed for 48 hours. The patients were again examined under sedation in the operation room for further evaluation six months after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years old
2. Occurrence of complex perianal fistula
3. Informed consent

Exclusion Criteria:

1. Active inflammatory bowel disease
2. Synchronous perianal abscess
3. Alcohol,narcotic and stimulant consumption
4. Having active Hepatitis B,C,HIV or TB
5. Peregnancy and lactation
6. Uncontrolled diabetes mellitus
7. Evidence of surgical contraindication
8. Psychological disorders and noncooperative patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Safety of injected exosomes | 3 months
  assessing the adverse outcomes after an injection such as acute allergic reactions, systemic effects such as fever, tachycardia, nausea and vomiting, diarrhea, cardinal manifestations, neutropenia, leukopenia, hemolysis, and local reactions such as cellulitis, abscess, skin rash, bleeding, necrosis
clinical Efficacy of injected exosomes | 3 months
  They are assessing the clinical response to therapy which might demonstrate the closure of refractory fistulas. These results include a full fistula closure in clinical observation and radiological assessments by MRI. Clinical improvement can be described as improvements in clinical manifestations such as pain, discharge, and bloody discharges. The fistulae are also assessed with MRI scans.
inflammatory markers | 3 months
  assessing inflammatory markers through laboratory workup, including CRP, IL-6, TNF-a, calprotectin

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Colorectal Surgery, Department of Surgery, Tehran University of Medical Sciences, Tehran, Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided